CLINICAL TRIAL: NCT05249699
Title: The Prophylaxis of Tuberculosis According to TSPOT Results After Kidney Transplantation (PTTKT):Protocol for an Open-label, Prospective, Randomized, 3-arm, Controlled Trial
Brief Title: The Prophylaxis of Tuberculosis According to TSPOT Results After Kidney Transplantation
Acronym: PTTKT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Tao Lin, Professor Tao Lin, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WestChinaH-PTTKT
Record Dates: First submitted 2021-10-19; First posted 2022-02-22 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Kidney Transplant Infection; Tuberculosis; Isoniazid Toxicity
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive TSPOT results with clinical risk factors group (Experimental): patients receive isoniazid 300mg once daily for six months after kidney transplant surgery form discharge
  Interventions: Drug: Isoniazid
- Negative TSPOT results with clinical risk factors group (Placebo Comparator): patients receive no additional therapy
  Interventions: Other: without any additional anti-tuberculosis treatment
- Clinical risk factors group (Experimental): patients receive isoniazid 300mg once daily for six months after kidney transplant surgery form discharge
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Isoniazid — prevent the development of tuberculosis
  Arms: Clinical risk factors group; Positive TSPOT results with clinical risk factors group
Other: without any additional anti-tuberculosis treatment — reduce the number of Participants With Treatment-Related Adverse Events
  Arms: Negative TSPOT results with clinical risk factors group

SUMMARY:
Organ transplant recipients are a high incidence group of tuberculosis infection, and the incidence rate is 7-27 times that of the general population. The prevention of postoperative tuberculosis infection is an important part of kidney transplant recipients postoperative follow-up. Taking reasonable tuberculosis prevention strategies for organ transplant recipients can better prevent the occurrence of postoperative tuberculosis and reduce the unreasonable use of anti-tuberculosis drugs. The previous screening methods for active tuberculosis mainly include sputum smear culture, tissue biopsy, tuberculin skin test, tuberculosis antibody, tuberculosis DNA, and chest imaging. However, there is still a lack of accurate and effective means for screening for latent tuberculosis infection. The tuberculosis interferon-γ release test has recently received more and more attention as a means of screening for potential tuberculosis infection. However, how to apply tuberculosis interferon-γ release test in clinical practice is still controversial. The investigators hope to explore the clinical application prospects and practical value of tuberculosis interferon-γ release test through this research.

According to the conclusion of the retrospective study, the investigators found that the recipients with negative TSPOT result maybe don't need follow the isoniazid treatment to prevent the development of tuberculosis even though participants have clinical risk factor of tuberculosis(include past tuberculosis history, the close contact with active tuberculosis patients, an area with a high incidence of tuberculosis, abnormal chest x ray performance ).

The investigators will divided the recipients with tuberculosis risk factors into three groups randomly. Of course, the invention require written informed consent. The first group with positive tuberculosis interferon gamma release assay (TSPOT) result will follow through with the treatment ,which is a daily dose of isoniazid for six months(300mg daily) after kidney transplant surgery. The second group with negative TSPOT result will not follow through the isoniazid treatment. The third group will follow through with the isoniazid treatment no matter their TSPOT results. The investigators will conduct a prospective clinical trial with the first aim of exploring the effectiveness of TSPOT results in kidney transplant recipients with clinical tuberculosis risk factors, and the second aim of exploring the benefit of the isoniazid treatment follow the TSPOT results rather than clinical risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. living-donor kidney transplantation;
2. eGFR level > 45ml/min/1.73m2 at discharge;
3. 18<Age <65years;
4. receiving standard triad immunosuppressive regimen

Exclusion Criteria:

1. alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 or more of upper limit of normal
2. Combined with HBV/HCV/HIV/TB infection in the donor or recipient;
3. Malignancy history in the donor and recipient;
4. organ transplant history in the recipient.
5. The positive TSPOT result or past TB history in the donor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the incidence of tuberculosis in these groups. | 12 months
  The primary objective of this study is to evaluate the incidence of tuberculosis between these groups. The incidence of tuberculosis was assessed by WHO TB guidelines 2021.

SECONDARY OUTCOMES:
The secondary outcome is subject incidence of adverse events | 12 months
  The primary objective of this study is to evaluate the safety of isoniazide among the kidney transplant recipients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim H, Kim SH, Jung JH, Kim MJ, Kim H, Shin S, Chong YP, Kim YH, Lee SO, Choi SH, Kim YS, Woo JH, Park SK, Han DJ. The usefulness of quantitative interferon-gamma releasing assay response for predicting active tuberculosis in kidney transplant recipients: A quasi-experimental study. J Infect. 2020 Sep;81(3):403-410. doi: 10.1016/j.jinf.2020.06.070. Epub 2020 Jun 29. PMID 32610111
- [Background] Shu CC, Tsai MK, Lin SW, Wang JY, Yu CJ, Lee CY. Latent Tuberculosis Infection Increases in Kidney Transplantation Recipients Compared With Transplantation Candidates: A Neglected Perspective in Tuberculosis Control. Clin Infect Dis. 2020 Aug 14;71(4):914-923. doi: 10.1093/cid/ciz851. PMID 32620949
- [Background] Kim SH, Lee SO, Park IA, Kim SM, Park SJ, Yun SC, Jung JH, Shin S, Kim YH, Choi SH, Kim YS, Woo JH, Park SK, Park JS, Han DJ. Isoniazid treatment to prevent TB in kidney and pancreas transplant recipients based on an interferon-gamma-releasing assay: an exploratory randomized controlled trial. J Antimicrob Chemother. 2015 May;70(5):1567-72. doi: 10.1093/jac/dku562. Epub 2015 Jan 20. PMID 25608587
- [Background] Kim SH, Lee SO, Park JB, Park IA, Park SJ, Yun SC, Jung JH, Kim YH, Kim SC, Choi SH, Jeong JY, Kim YS, Woo JH, Park SK, Park JS, Han DJ. A prospective longitudinal study evaluating the usefulness of a T-cell-based assay for latent tuberculosis infection in kidney transplant recipients. Am J Transplant. 2011 Sep;11(9):1927-35. doi: 10.1111/j.1600-6143.2011.03625.x. Epub 2011 Jul 12. PMID 21749641